CLINICAL TRIAL: NCT01574833
Title: Phase 4 Study of Early Applied Pulsed Electromagnetic Field in the Treatment of Postoperative Delayed Union of Long-bone Fractures
Brief Title: Early Application of Pulsed Electromagnetic Field in the Treatment of Postoperative Delayed Union
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jin XIONG, Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QYK10147
Record Dates: First submitted 2012-04-07; First posted 2012-04-10 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Fracture; Delayed Union of Fracture
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEMF (Active Comparator): arm that receive PEMF treatment
  Interventions: Device: pulsed electromagnetic field
- Sham (Sham Comparator): arm that receive sham treatment
  Interventions: Device: sham

INTERVENTIONS:
Device: pulsed electromagnetic field — PEMF treatment
  Arms: PEMF
Device: sham — sham treatment
  Arms: Sham

SUMMARY:
The investigators hypothesized that early applied pulsed electromagnetic field treatment on delayed union might lead to increased rate of fracture union and shortened period of treatment.

ELIGIBILITY:
Inclusion Criteria:

* The failure of healing after at least 16 weeks and not more than 9 months following surgical reduction and fixation of the fracture.

Exclusion Criteria:

* Implant loosening or failure, infection, established nonunion, fracture gap greater than 5 mm, presence of implant within the fracture gap, metabolic disorders or received medication affecting fracture healing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-03; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
percentage of patient achieving fracture union | 12 months

SECONDARY OUTCOMES:
pain | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China